CLINICAL TRIAL: NCT04454385
Title: The Correlations of FeNO, Blood Eosinophils and Lung Function in Well-controlled Asthma Based on Asthma Controlled Questionnaires
Brief Title: The Correlations of FeNO, Blood Eosinophils and Lung Function in Well-controlled Asthma
Status: Completed | Type: Observational
Sponsor: Hat Yai Medical Education Center (Other)
Responsible Party: Principal Investigator, Narongwit Nakwan, Asst.prof Narongwit Nakwan, Hat Yai Medical Education Center
Other Study IDs: 56/2563
Record Dates: First submitted 2020-06-28; First posted 2020-07-01 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-06

CONDITIONS: Asthma
Keywords: FeNO; Blood eosinophil; Pulmonary function test; Well controlled asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood for CBC analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Patients with well controlled asthma — Patients with well controlled asthma
  The following parameters are to be evaluated:
  Blood eosinophils FeNO Findings on lung function test

SUMMARY:
In Asthma, the levels of exhaled FeNO is correlated to sputum eosinophils particularly in the patient with poor controlled asthma or severe asthma. Moreover, the blood eosinophils had been studied that are also correlated to sputum eosinophils in similar patients group. According to well controlled asthma, althoug hin clinical practice guidelines recommend that the stepping down therapy should be considered to those patients due to the risks or costs of daily treatment, there is previous study has been shown that the airway hyperresponsiveness and sputum eosinophilia are predictors of loss of control during dose reduction. And, these tests are not readily available in primary care. However, there is limit number of clinical study to study the correlation of biologic markers among the patients with well controlled level before the stepping down management.

DETAILED DESCRIPTION:
This is a single prospective trial. Enrollment will continue until 50 patients with well controlled asthma have been entered into this trial and have completed blood tests and spirometry. In this trial, the following parameters are to be evaluated:

Blood eosinophils (absolute and relative) FeNO Pulmonary lung function test: FEV1, FVC, PF, MMEF 25-75%, % reversibility

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of asthma (according to the guidelines)
* Age >15 years
* Patients with treating with step 3 base on GINA by only low dose ICS/LABA without oral bronchodilator with being in well controlled asthma based on ACT (> = 23) and ACQ-7 (<0.75) for at least 12 weeks
* Ability to provide informed consent and do spirometry following ATS guideline

Exclusion Criteria:

* Pulmonary infection or exacerbation within the last 12 weeks before enrolment
* Patients with preceding taken systemic steroid 12 week before enrolment
* Additional pulmonary diseases (pneumonia, lung cancer, tuberculosis, interstitial lung disease)
* A history of smoking >= 10 pack-year

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with well controlled asthma treating with step 3 base on GINA by only low dose ICS/LABA based on ACT (> = 23) and ACQ-7 (<0.75) for at least 12 weeks
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Assessment of eosinophilic inflammation by correlating blood eosinophil count, FeNO measurement and lung function test | 3 months
  Correlation of FeNO, blood eosinophils, lung function test in patients with well controlled asthma before stepping down medication

CONTACTS AND LOCATIONS:
Locations (1):
- Narongwit Nakwan, Hat Yai, Changwat Songkhla, Thailand